CLINICAL TRIAL: NCT05028478
Title: An Open-Label, Multi-center, Phase I/II Study of CN202 in Adult Subjects With Locally Advanced or Metastatic Solid Tumors or Hematologic Malignancies
Brief Title: A Study of CN202 in Adult Subjects With Locally Advanced or Metastatic Solid Tumors or Hematologic Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Curon Biopharmaceutical (Australia) Co Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN202-102
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor; Hematologic Malignancies
MeSH Terms: conditions — Neoplasm Metastasis; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Four planned CN202 dose level of 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg
  Subjects will receive CN202 by intravenous infusion (IV) on Day 1 of each cycle (once every 2 weeks) for up to 24 months
  Interventions: Drug: CN202

INTERVENTIONS:
Drug: CN202 — Participants will receive CN202 by IV infusion on Day 1 of each cycle (once every 2 weeks). The 4 planned dose levels are 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg

SUMMARY:
The study is designed to evaluate the safety, tolerability, pharmacokinetic characteristics and anti-tumor activity of CN202 in adult subjects with locally advanced or metastatic solid tumor or hematologic malignancies

DETAILED DESCRIPTION:
This is a multi-centre, open-label, Phase I/II study in adult subjects with locally advanced or metastatic solid tumor or hematologic malignancies.

The study consists of three parts

Phase Ia: Dose Escalation: This is a dose escalation for assessment of dose-limiting toxicities (DLT) at approximately four dose levels in subjects with locally advanced or metastatic solid tumor or hematologic malignancies.

Phase Ib: Dose Expansion: To evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of CN202, prior to determination of Maximum tolerated dose (MTD)

Phase II: To further evaluate the safety, tolerance, pharmacokinetic characteristics, and anti-tumor activity of CN202 in subjects with select tumors. All subjects will receive the recommended Phase II dose of CN202.

There will be 13 to 24 subjects enrolled in phase Ia, 12 to 40 subjects in phase Ib and 15 to 100 subjects in phase II

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ age of 18 on the day of signing informed consent;
2. Histologically or cytologically diagnosed metastatic or locally advanced solid tumor or hematologic malignancy (unresectable), for whom no effective standard anti-tumor therapy existed or in the opinion of the Investigator have been considered ineligible for standard anti-tumor therapy at this stage, or are intolerant to standard anti-tumor therapy, or standard therapy had failed or the subject has refused standard anti-tumor therapy, or recurrent and progressing since last line anti-tumor therapy;
3. Representative tumor specimens in paraffin blocks (preferred) or at least 10 unstained slides, with an associated pathology report, requested at any time prior to study entry. Only tissue from core needle, punch, or excisional biopsy sample collection will be accepted. If archival tissue is insufficient or unavailable, the subjects may still be eligible upon discussion with Medical Monitor and approved by sponsor.
4. At least 1evaluable tumor lesion per RECIST v1.1 (Solid Tumors) and Lugano 2014 Criteria (Lymphoma). Disease-specific criteria will be used for prostate cancer and or other tumors. The subjects enrolled in phase Ib/II study must have measurable disease.
5. Subjects with Eastern Cooperative Oncology Group (ECOG) performance score of 0 to1;
6. At least 3 months of expected survival;
7. Female subjects must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception method from Screening until the end of the Safety Follow-up period, 90 (±7 days) days after the last dose of the study drug. Double contraception is defined as a condom AND one other from of the following:

   1. Established hormonal contraception (with approved OCPs, long-acting implantable hormones, injectable hormones);
   2. A vaginal ring or an intrauterine device (IUD);
   3. Documented evidence of surgical sterilization at least 6 months prior to screening (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner).
   4. Women not of childbearing potential must be post-menopausal for ≥12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/L at Screening for amenorrhoeic female participants. Females who are abstinent from heterosexual intercourse will also be eligible.
   5. Periodic abstinence (eg, calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not considered highly effective methods of birth control. Participant complete abstinence for the duration of the study and for 1 month after the last study treatment is acceptable.
   6. Female participants who are in same-sex relationships are not required to use contraception.

   Male subjects willing to use a highly effective method of contraception throughout the study period and for 90 days after the last dose of study drug.
8. Subjects must be able to understand and sign the paper informed consent before any study specific procedure.

Exclusion Criteria:

1. Received anti-tumor therapy, including radiotherapy, chemotherapy, hormonal therapy, immunotherapy, within 3 weeks prior to initiation of study treatment, however, the following are allowed:

   * Palliative radiation therapy > 2 weeks.
   * Small molecule targeted therapy > 2 weeks. But subject who has had anti-EGFR or anti-TKI (egerlotinib, gefitinib, afatinib, or crizotinib) > 1 week prior to the first dose of study therapy.
   * Use of immunomodulatory drugs > 14 days or 5 half-lives of the drug prior to the first dose of study drug (whichever is shorter), including but not limited to thymosin, interleukin-2 (IL-2), interferon (IFN), etc.
   * Herbal therapy > 1 week.
   * Hormone-replacement therapy or oral contraceptives.
   * Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists or antagonists for prostate cancer.
2. The subjects had prior treatment with anti-PD-L1 or anti-PD-1 therapeutic antibody, with the following exceptions:

   1. The subjects can be enrolled in Phase Ia study if no history of severe immune-related adverse effects from checkpoint inhibitor treatment or any that has led to discontinuation (CTCAE Grade 3 and 4).
   2. The subjects may be enrolled in Phase Ib/II study if the following requirements are met:

      * > 6 weeks from the last dose of anti-PD-L1 or anti-PD-1 therapeutic antibody
      * No history of severe immune-related adverse effects from checkpoint inhibitor treatment or any that has led to discontinuation (CTCAE Grade 3 and 4).
      * at least 3 months on PD1 with evidence of benefit or stable disease as per investigator' judgment.
3. Subjects who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

   * > 6 weeks from the last dose of anti-CTLA-4
   * No history of severe immune-related adverse effects from anti-CTLA-4 (CTCAE Grade 3 and 4)
4. Received other investigational agents (not yet approved by any regulatory agency) within 4 weeks prior to the first dose of study drug;
5. Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks prior to the first dose of study drug, or elective surgery during the trial;
6. Systemic application of corticosteroids (prednisone > 10 mg/day or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of study drug;

   • Exceptions: topical, ocular, intra-articular, intranasal, inhaled corticosteroids, or short-term corticosteroids for prophylaxis (eg, contrast allergy prophylaxis).
7. Use of live attenuated vaccine within 4 weeks prior to the first dose of study drug;

   * Exception: Approved COVID-19 vaccine is allowed, but the last dose of COVID-19 vaccine should be administered 2 weeks prior to first dose of study drug;
   * For active subjects enrolled in this study, COVID-19 vaccination is allowed after 8 weeks treatment have been completed and the safety data have been obtained to make conclusion regarding the safety of the investigational product.
8. Adverse reactions prior to anti-tumor therapy that have not recovered to ≤ Grade 1 assessed by CTCAE Version 5.0 (except for toxicities such as alopecia judged by the Investigator as no safety risk);
9. Clinically symptomatic metastases to the central nervous system (CNS) or meninges, or other evidence of uncontrolled metastases to the CNS or meninges of the subject, judged by the Investigator. Subjects are eligible if metastases have been treated, subjects are neurologically stable for at least four weeks and not requiring steroid therapy for at least one week prior to Cycle 1 Day 1.
10. Active infection and in current need of, or likely to need, intravenous anti-infective therapy;
11. History of immunodeficiency, including history of any positive test result for human immunodeficiency virus (HIV) antibody;
12. Active hepatitis B or hepatitis C infection: defined as having a positive hepatitis B surface antigen (HBsAg) test and/or detectable level of HBV DNA at Screening or hepatitis C infection defined as having a positive HCV antibody test followed by a positive HCV RNA test at Screening. HCV negative subjects are allowed to enrol. But in Phase Ib/II, the subjects with HBsAg+ but HBV DNA negative are allowed to be enrolled in HCC cohort with the use of antiviral therapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-10-22 (Estimated); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-10-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CN202 administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies through adverse events as assessed by NCI-CTCAE v5.0 | Measurements at Baseline till 90 days after the last dose of study drug
  Number of participants with treatment related adverse events as assessed by NCI-CTCAE v5.0
To evaluate the dose-limiting toxicity (DLT) and to determine the maximum tolerated dose (MTD) of CN202 when administered as a single-agent to subjects | DLT assessed within 21 days after the first dose of CN202
  Measured by Incidence of dose limiting toxicities (DLT) during the first cycle of treatment and DLT observation period
To identify a recommended Phase II dose (RP2D) of CN202 | Baseline to End of the Treatment assessed up to an average of 24 months
  The recommended Phase II dose (RP2D) will be determined based on safety, efficacy, pharmacokinetics and pharmacodynamic date of CN202
To evaluate the anti-tumor activity of CN202 in selected solid tumors or hematologic malignancies as determined by Objective Response Rate (ORR) | Baseline to End of the Treatment assessed up to an average of 24 months
  Measured/determined by Objective Response Rate

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of CN202 administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies through Electrocardiogram (ECG) | Baseline to End of the Treatment assessed up to an average of 24 months
  Measured by ECG as assessed by the P wave, the QRS complex, and T wave
To evaluate the safety and tolerability of CN202 administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies through vital signs as assessed by heart rate | Baseline to End of the Treatment assessed up to an average of 24 months
To evaluate the safety and tolerability of CN202 administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies through vital signs as assessed by body temperature | Baseline to End of the Treatment assessed up to an average of 24 months
To evaluate the safety and tolerability of CN202 administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies through vital signs as assessed by pulse, systolic blood pressure, and diastolic blood pressure | Baseline to End of the Treatment assessed up to an average of 24 months
To evaluate the safety and tolerability of CN202 administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies through vital signs as assessed by respiratory rate | Baseline to End of the Treatment assessed up to an average of 24 months
To evaluate the pharmacokinetic (PK) of CN202 when administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies | Baseline to End of the Treatment assessed up to an average of 24 months
  The following parameter is used for evaluation during PK assessments: maximum concentration (Cmax)
To evaluate the pharmacokinetic (PK) of CN202 when administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies | Baseline to End of the Treatment assessed up to an average of 24 months
  The following parameter is used for evaluation during PK assessments: area under the concentration-time curve (AUC)
To evaluate the pharmacokinetic (PK) of CN202 when administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies | Baseline to End of the Treatment assessed up to an average of 24 months
  The following parameter is used for evaluation during PK assessments: half-life (t½)
To assess the immunogenic potential of CN202 by measuring anti-CN202 antibodies through Immunogenicity analysis test results | Baseline to End of the Treatment assessed up to an average of 24 months
  Measured through immunogenicity analysis test results (anti-drug antibodies and Neutralizing antibodies) and days from first dosing to positive result of anti-drug antibodies (ADA) or Neutralizing antibodies (NAb)
To assess the pharmacodynamic (PD) of CN202 when administered to subjects with locally advanced or metastatic solid tumor or hematologic malignancies | Baseline to End of the Treatment assessed up to an average of 24 months
  The pharmacodynamic profile assessed based on the analysis of PD-L1 receptor occupancy (RO) and biomarkers in peripheral blood and tumor tissues

CONTACTS AND LOCATIONS:
Overall Officials: Gary Richardson, Principal Investigator — Cabrini Oncology Research; Morteza Aghmesheh, Principal Investigator — Southern Medical Day Care Centre